CLINICAL TRIAL: NCT03865420
Title: Amyotrophic Lateral Sclerosis (ALS) Families Project
Status: Recruiting | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Other Study IDs: AAAR7275
Record Dates: First submitted 2019-02-25; First posted 2019-03-06 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: ALS
Keywords: Pre-symptomatic; Familial; FALS; Genetic testing; C9orf72; SOD1; TARDBP; FUS; VCP; PFN1
MeSH Terms: conditions — Frontotemporal Dementia With Motor Neuron Disease

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA, RNA, spinal fluid, plasma, serum and Peripheral blood mononuclear cells (PBMCs)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This program provides family members of individuals with familial ALS the opportunity to contribute to research focused on learning more about why motor neuron degeneration begins and how or why it progresses. This study provides genetic counseling and testing to help participants understand and manage their risk and determine if they want to learn their genetic status. This study will follow unaffected ALS gene mutation carriers on an annual basis to gather essential information that will ultimately help researchers develop novel therapies for the prevention and treatment of ALS.

DETAILED DESCRIPTION:
Approximately 10% of people with amyotrophic lateral sclerosis (ALS), or Lou Gehrig's Disease, have a family history of ALS or a related condition called frontotemporal dementia (FTD). In most of these familial cases, and a significant number of "sporadic" patients with no family history, a mutation is present in one of a growing number of genes that have been associated with ALS and/or FTD.

The ALS Families Project will study unaffected carriers of ALS/FTD-associated gene mutations to investigate the first steps in the disease process that leads to motor neuron degeneration, with the goal of identifying early disease targets and points of intervention to slow or stop disease onset and progression.

Unaffected individuals who have either a family member with a known ALS/FTD-associated gene mutation or have a strong family history of ALS and FTD are invited to participate in the ALS Families Project. For those who enroll, research visits will occur every 6-12 months.

ELIGIBILITY:
Inclusion Criteria:

* Men or women of any race or ethnicity aged 18 or older
* No symptoms of ALS or fronto-temporal dementia at enrollment
* Scenario 1: has already had genetic testing that identified an ALS-spectrum gene mutation.
* Scenario 2: has a first degree relative who was/is an obligate carrier of a familial ALS-spectrum gene mutation.
* Scenario 3: has a first degree relative who has/had an ALS-spectrum diagnosis who had a confirmed ALS-spectrum gene mutation or comes from a family with a high burden of ALS-spectrum diagnoses and a known ALS-spectrum gene mutation.
* Scenario 4: is deemed to be at high risk for carrying an ALS-spectrum gene mutation as judged by a review of the family structure and genetic information by the study team.
* Willing to undergo genetic analysis, with option of whether or not to learn results
* Willing to travel to Columbia University Irving Medical Center (CUIMC) every 6-24 months for study procedures
* Capable of providing informed consent and following study procedures, or has a legally authorized representative who is able to consent for the subject.

Exclusion Criteria for participation in biosample portion of the study:

* Known HIV
* Known hepatitis B
* Known hepatitis C

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Unaffected individuals who have either a family member with a known ALS/FTD-associated gene mutation or have a strong family history of ALS and FTD.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-09-11 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Time to emergence of symptoms attributable to gene mutations | Up to 10 years
  Emergence of symptoms will defined by the development of any of the following: a) any weakness on neurological examination, b) evidence of nerve loss on electromyography (EMG)-nerve conduction studies, or c) evidence of cognitive impairment on the ECAS or ALS-Cognitive Behavioral Scale (ALS-CBS).

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Harms, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No